CLINICAL TRIAL: NCT02145845
Title: Pilot Safety Study of Injectable Small Intestine Submucosa (SIS) for Critical Limb Ischemia
Brief Title: Pilot Safety Study of Injectable SIS for Critical Limb Ischemia
Acronym: CLIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-013
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: critical limb ischemia; wound healing; amputation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Injectable SIS
  Interventions: Device: Injectable SIS

INTERVENTIONS:
Device: Injectable SIS — Injectable SIS

SUMMARY:
This study is intended to collect safety and effectiveness data on the Cook Injectable Small Intestinal Submucosa (SIS)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of critical limb ischemia
* Rutherford 4-5 or Leriche-Fontaine IIIB
* Patient unable to be treated by endovascular or surgical means

Exclusion Criteria:

* Patient's age is <21
* Patient is pregnant or breast-feeding (or is planning to become pregnant within the next year)
* Patient has had a previous surgery, within 30 days of the study procedure
* Patient has any planned surgical or interventional procedure within 30 days after the study procedure
* Patient has a life expectancy less than 1 year
* Patient has a known allergy to pigs or pig products, or has a religious or cultural objection to the use of pig tissue
* Additional restrictions as specified in the Clinical Investigation Plan

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2017-06-05 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Frequency and types of adverse events after treatment with the Cook Injectable SIS | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Vaclav Prochazka, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia